CLINICAL TRIAL: NCT02359045
Title: A Randomized, Open-label, Single-center, Cross-over Study in Healthy Subjects to Assess the Relative Bioavailability of EPA and DHA Delivered by Three New Capsule Formulation Prototypes in Relation to the Current Epanova® Capsule Under Fasting (Part 1) and Fed (Part 2) Conditions
Brief Title: Study in Healthy Subjects to Compare the Concentrations of the Omega-3 Fatty Acids EPA and DHA in Blood When Delivered as Three New Capsules in Relation to the Epanova® Capsule Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5884C00003
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Relative Bioavailability; AUC; Cmax; Pharmacokinetics
Keywords: Omega-3-carboxylic acids,; Phase I,; Healthy Subjects,; Pharmacokinetics,; Relative bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Treatment A-B-C-D (Experimental): Subjects received a single dose of D1400147 (Treatment A: Omega-3-carboxylic acids 2000 mg uncoated capsules), D14000136 (Treatment B: Omega-3-carboxylic acids 2000 mg coated capsules coat 1), D14000137 (Treatment C: Omega-3-carboxylic acids 2000 mg coated capsules coat 2) and Epanova® (Treatment D: Epanova capsules 1000 mg) under fasted condition.
  Interventions: Drug: D1400147; Drug: D14000136; Drug: D14000137; Drug: Epanova®
- Part 2: Treatment A-B/C-D (Experimental): Subjects received a single dose of D1400147 (Treatment A: Omega-3-carboxylic acids 2000 mg uncoated capsules), D14000136 (Treatment B: Omega-3-carboxylic acids 2000 mg coated capsules coat 1) or D14000137 (Treatment C: Omega-3-carboxylic acids 2000 mg coated capsules coat 2) and Epanova® (Treatment D: Epanova capsules 1000 mg) under fed condition.
  Interventions: Drug: D1400147; Drug: D14000136; Drug: D14000137; Drug: Epanova®

INTERVENTIONS:
Drug: D1400147 — Treatment A
Drug: D14000136 — Treatment B
Drug: D14000137 — Treatment C
Drug: Epanova® — Treatment D

SUMMARY:
This study is a randomized, open-label, cross-over study in healthy subjects performed at a single study center. The study is divided into two parts, Part 1 and Part 2. The purpose of the study is to compare the pharmacokinetics (PK) of three different prototype capsule formulations (omega-3-carboxylic acids test formulations) with Epanova® capsules 1000 mg under fasted conditions in Part 1 and under fed conditions in Part 2. The results will be used as basis for choice of formulation for further pharmaceutical development.

DETAILED DESCRIPTION:
To assess the relative bioavailability of the different omega-3-carboxylic acids prototype capsule formulations in relation to Epanova® capsules 1000 mg under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures.
* Healthy male and female (non-childbearing potential) subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the clinical unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  * Post-menopausal, defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments, and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy or tubal ligation.
* Have a body mass index (BMI) between 18.5 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influences the results or the potential subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* Consumption of poppy seeds within 7 days of first administration of IMP.
* Consumption of fish within 7 days prior to admission to the clinical unit.
* Used fish oil, other omega-3 fatty acids (EPA and/or DHA) containing supplements within 1 month of admission to the clinical unit.
* Have a known sensitivity or allergy to soybeans, fish and/or shellfish.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2015-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore, 3001 S. Hanover St., Baltimore, MD 21225, United States of America
Locations (1):
- Research Site, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Baltimore, USA. All enrolled participants were included in the study.
  A total of 137 participants were enrolled (signed ICF) and underwent screening visits, out of which 55 were screen failures and 82 were independently enrolled in the study.
Pre-assignment Details: All the randomized participants were divided into 2 parts. Part 1- 4 sequence for 4 periods, 4 treatments: (ADBC, BACD, CBDA, DCAB) A- D1400147, B- D14000136, C- D14000137 & D- Epanova.
  Part 2- 6 sequence for 3 treatments, 3 periods: (ABC, BCA, CAB, ACB, BAC, CBA) A-D1400147, B- D14000136 or D14000137 & C- Epanova.
Groups:
- Part 1: Subjects received a single dose of 4 treatments for 4 periods to assess the relative bioavailability and to characterize and compare the PK profiles of the three different prototype capsule formulations (Treatment A, B, C) in relation to Epanova capsules (Treatment D), under fasted conditions.
  A- D1400147, B- D14000136, C- D14000137 & D- Epanova.
- Part 2: Subjects received a single dose of 3 treatments for 3 periods to assess the relative bioavailability and to characterize and compare the PK profiles of the two different prototype capsule formulations (Treatment A, B) in relation to Epanova capsules (Treatment C), under fed conditions.
  A-D1400147, B- D14000136 or D14000137 & C- Epanova.
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 40 | 42
Completed | 36 | 39
Not Completed | 4 | 3
Not completed — Eligibility criteria not fulfilled | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (9.97) | 37.1 (9.97) | 37.9 (9.97)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 0 | 5 | 5
  Male | 40 | 37 | 77

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC) Assessed for Eicosapentaenoic Acid (EPA) After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: Subjects were analyzed based on PK analysis set. It consisted of all subjects in the safety analysis set for whom the primary PK parameters could be calculated for at least 2 treatment periods including the reference formulation, and who had no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Groups:
- Treatment A_Part 1: Subjects received a single dose of Treatment A (D1400147: Omega-3-carboxylic acids 2000 mg uncoated capsules) under fasted condition.
- Treatment B_Part 1: Subjects received a single dose of Treatment B (D14000136: Omega-3-carboxylic acids 2000 mg coated capsules coat 1) under fasted condition.
- Treatment C_Part 1: Subjects received a single dose of Treatment C (D14000137: Omega-3-carboxylic acids 2000 mg coated capsules coat 2) under fasted conditions.
- Treatment D_Part 1: Subjects received a single dose of Treatment D (Epanova capsules 1000 mg) under fasted conditions.
- Treatment A_Part 2: Subjects received a single dose of Treatment A (D1400147: Omega-3-carboxylic acids 2000 mg uncoated capsules) under fed conditions.
- Treatment B_Part 2: Subjects received a single dose of Treatment B as D14000136: Omega-3-carboxylic acids 2000 mg coated capsules coat 1 or D14000137: Omega-3-carboxylic acids 2000 mg coated capsules coat 2, under fed conditions.
- Treatment C_Part 2: Subjects received a single dose of Treatment C (Epanova capsules 1000 mg) under fed conditions.
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 34 | 28 | 24 | 30 | 36 | 38 | 39
µg*h/mL | 2010 (47.9) | 1400 (88.6) | 744 (81.5) | 1720 (54.5) | 3460 (34.0) | 3010 (34.7) | 3450 (33.7)

2. Primary Outcome: AUC Assessed for Docosahexaenoic Acids (DHA) After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg*h/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 3 | 8 | 2
(μg*h/mL) | 783 (72.6) | 502 (78.4) | 399 (106) | 674 (38.4) | 791 (40.4) | 501 (79.1) | 325 (15.8)

3. Primary Outcome: AUC Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol*hr/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 22 | 15 | 13 | 15 | 19 | 21 | 21
(nmol*hr/mL) | 10400 (52.3) | 6870 (72.7) | 4250 (102) | 7710 (92.6) | 15300 (47.6) | 12500 (43.8) | 15800 (50.6)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 72 Hours After Dosing {AUC(0-72)} Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (0-72) for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg*h/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 35 | 36 | 39 | 40 | 40
(μg*h/mL) | 1680 (37.5) | 1080 (74.4) | 564 (93.8) | 1080 (88.4) | 2570 (27.8) | 2310 (27.5) | 2620 (28.4)

5. Primary Outcome: AUC (0-72) Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (0-72) for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg*h/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 35 | 35 | 38 | 39 | 40
(μg*h/mL) | 577 (65.7) | 405 (78.5) | 309 (92.0) | 339 (135) | 610 (57.0) | 483 (53.4) | 531 (55.6)

6. Primary Outcome: AUC (0-72) Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (0-72) for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol*hr/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(nmol*hr/mL) | 7200 (44.0) | 4560 (80.5) | 2710 (92.3) | 4470 (96.9) | 10200 (31.3) | 9030 (28.2) | 10100 (32.1)

7. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of Cmax for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg/mL) | 93.5 (46.5) | 54.5 (94.8) | 24.8 (98.1) | 50.0 (108) | 140 (41.4) | 119 (38.2) | 156 (40.3)

8. Primary Outcome: Cmax Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of Cmax for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg/mL) | 46.7 (44.9) | 31.6 (67.7) | 19.0 (67.7) | 24.0 (83.0) | 55.4 (46.3) | 45.3 (41.8) | 58.0 (50.7)

9. Primary Outcome: Cmax Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of Cmax for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(nmol/mL) | 447 (46.2) | 276 (84.0) | 139 (84.4) | 241 (91.4) | 626 (42.1) | 522 (39.9) | 690 (42.0)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Analyte Concentration {AUC (Last)} Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (last) for EPA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentration.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg*h/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg*h/mL)
  EPA (Baseline Subtracted) | 1670 (37.7) | 1080 (74.9) | 518 (116) | 1080 (89.1) | 2570 (27.9) | 2310 (27.4) | 2620 (28.5)
  EPA (Baseline Unadjusted) | 2800 (31.0) | 2190 (41.8) | 1620 (42.6) | 2150 (44.9) | 3730 (27.3) | 3500 (24.8) | 3850 (25.2)

11. Secondary Outcome: AUC (Last) Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (last) for DHA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentration.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg*h/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg*h/mL)
  DHA (Baseline Subtracted) | 553 (72.3) | 391 (83.3) | 286 (98.5) | 328 (142) | 588 (60.2) | 484 (57.7) | 527 (58.2)
  DHA (Baseline Unadjusted) | 4770 (22.2) | 4700 (24.4) | 4510 (19.3) | 4520 (20.8) | 5340 (28.4) | 5290 (26.0) | 5360 (27.7)

12. Secondary Outcome: AUC (Last) Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of AUC (last) for Total (combined) EPA + DHA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentration.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol*hr/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(nmol*hr/mL)
  Total (combined) EPA + DHA(Baseline Subtracted) | 7180 (44.5) | 4540 (81.4) | 2570 (100) | 4340 (112) | 10200 (31.4) | 9040 (28.2) | 10200 (32.1)
  Total (combined) EPA + DHA(Baseline Unadjusted) | 24000 (23.3) | 21800 (26.0) | 19400 (21.3) | 21200 (25.0) | 28800 (25.4) | 27900 (22.5) | 29300 (24.0)

13. Secondary Outcome: Baseline Concentration (C0) Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of C0 for EPA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg/mL)
  EPA (Baseline Subtracted) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  EPA (Baseline Unadjusted) | 13.7 (54.2) | 13.3 (40.3) | 13.2 (42.3) | 12.8 (38.8) | 14.8 (48.6) | 15.6 (38.3) | 15.9 (40.6)

14. Secondary Outcome: C0 Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of C0 for DHA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (μg/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(μg/mL)
  DHA (Baseline Subtracted) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  DHA (Baseline Unadjusted) | 57.2 (24.8) | 59.0 (26.4) | 58.0 (20.9) | 57.1 (22.7) | 65.8 (29.4) | 66.6 (26.9) | 66.7 (29.1)

15. Secondary Outcome: C0 Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of C0 for Total (combined) EPA + DHA on baseline subtracted plasma concentrations and baseline unadjusted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nmol/mL)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(nmol/mL)
  Total (combined) EPA + DHA (Baseline Subtracted) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Total (combined) EPA + DHA (Baseline Unadjusted) | 223 (27.8) | 225 (26.6) | 223 (21.8) | 218 (22.4) | 65.8 (29.4) | 66.6 (26.9) | 66.7 (29.1)

16. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz) Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of t½λz for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 34 | 28 | 24 | 30 | 36 | 38 | 39
(hour) | 25.3 (44.3) | 26.0 (49.3) | 23.1 (59.7) | 29.2 (39.4) | 33.8 (42.8) | 31.2 (39.2) | 33.1 (49.5)

17. Secondary Outcome: t½λz Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of t½λz for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 3 | 8 | 2
(hour) | 24.1 (88.7) | 18.8 (51.7) | 13.0 (85.6) | 22.5 (77.1) | 24.6 (50.3) | 18.4 (135) | 4.56 (737)

18. Secondary Outcome: t½λz Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of t½λz for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 22 | 15 | 13 | 15 | 19 | 21 | 21
(hour) | 30.4 (65.5) | 23.8 (70.1) | 19.1 (76.1) | 23.4 (82.1) | 33.9 (62.5) | 30.3 (67.3) | 40.7 (80.7)

19. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of tmax for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(hour) | 6.02 [5.00 to 9.00] | 7.50 [5.00 to 12.00] | 8.99 [5.98 to 36.0] | 7.50 [5.98 to 24] | 6.00 [2.0 to 12.0] | 6.02 [3.00 to 24.0] | 6.00 [4.00 to 12.0]

20. Secondary Outcome: Tmax Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of tmax for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(hour) | 6.00 [5.00 to 9.03] | 7.5 [2.00 to 12.0] | 7.50 [2.02 to 72.0] | 7.49 [3.95 to 24.0] | 5.98 [2.0 to 9.02] | 6.00 [3.00 to 72.1] | 5.49 [3.00 to 8.97]

21. Secondary Outcome: Tmax Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of tmax for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: (hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 39 | 40 | 40
(hour) | 6.02 [5.00 to 9.03] | 7.50 [2.00 to 12.00] | 7.50 [4.98 to 72.0] | 7.51 [5.00 to 24.0] | 6.00 [2.0 to 9.02] | 6.00 [3.00 to 8.98] | 6.00 [3.00 to 8.97]

22. Secondary Outcome: Terminal Elimination Rate Constant (λz ) Assessed for EPA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of λz for EPA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (1/hour)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 34 | 28 | 24 | 30 | 36 | 38 | 39
(1/hour) | 0.0274 (44.3) | 0.0267 (49.3) | 0.0301 (59.7) | 0.0237 (39.4) | 0.0205 (42.8) | 0.0222 (39.2) | 0.0209 (49.5)

23. Secondary Outcome: λz Assessed for DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of λz for DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (1/h)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 3 | 8 | 2
(1/h) | 0.0287 (88.7) | 0.0369 (51.7) | 0.0531 (85.6) | 0.0308 (77.1) | 0.0282 (50.3) | 0.0377 (135) | 0.152 (737)

24. Secondary Outcome: λz Assessed for Total (Combined) EPA + DHA After Administration of Test Formulation 1, 2 and 3 and Reference Formulation.
Description: To assess the rate and extent of absorption of omega-3-carboxylic acids following single-dose oral administration of test formulation 1, 2 and 3 (Omega-3-carboxylic acids 2000 mg uncoated/coated capsules) and reference formulation (Epanova 1000 mg) under fasted (Part 1) and fed condition (Part 2), by assessment of λz for Total (combined) EPA + DHA on baseline subtracted plasma concentrations.
Time Frame: Pre-dose: -12, -1 and 0 hours and Post-dose: 0.5, 1, 2, 3, 4, 5, 6, 7.5, 9, 12, 24, 36, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (1/h)
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 22 | 15 | 13 | 15 | 19 | 21 | 21
(1/h) | 0.0228 (65.5) | 0.0291 (70.1) | 0.0363 (76.1) | 0.0297 (82.1) | 0.0204 (62.5) | 0.0229 (67.3) | 0.0170 (80.7)

25. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Summary of Adverse Events
Description: To assess the safety summary of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: Subjects were analyzed based on safety analysis set. Safety Analysis Set is defined as All subjects who received at least one dose of IMP were included in the safety analysis for the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants
  Any AE | 8 | 7 | 4 | 5 | 3 | 3 | 3
  Any AE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuationof IP | 0 | 0 | 0 | 0 | 0 | 0 | 1

26. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects Who Had at Least One Adverse Event
Description: To assess the safety by analyzing the number of subjects with at least one adverse event after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing.
Population: as for outcome 25
Measure: Number; unit: Partcipants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Partcipants
  Eyelid Edema | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ocular Hyperemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Vision Blurred | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal Distension | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Abdominal Pain | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Abdominal Pain Upper | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Diarrhea | 2 | 2 | 1 | 2 | 0 | 0 | 1
  Dry Mouth | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Frequent Bowel Movements | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Dyspepsia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Flatulence | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Catheter Site Bruise | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Catheter Site Phlebitis | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Catheter Site Swelling | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Vessel Puncture Site Hematoma | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Hordeolum | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Dizziness | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Dysgeusia | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Headache | 2 | 1 | 0 | 1 | 1 | 0 | 0
  Presyncope | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Somnolence | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Rhinorrhea | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sneezing | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Epistaxis | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hepatic Enzyme Increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neck Pain | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Acne | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hematoma | 0 | 0 | 0 | 0 | 0 | 1 | 0

27. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant Blood Pressure
Description: To evaluate the safety by assessing the number of subjects with clinically significant blood pressure after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant Pulse
Description: To evaluate the safety by assessing the number of subjects with clinically significant pulse after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant 12-lead Electrocardiograms (ECGs)
Description: To evaluate the safety by assessing the number of subjects with clinically significant 12-lead ECGs after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 39 | 39 | 37 | 37 | 37 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant Hematology Parameters
Description: To evaluate the safety by assessing the number of subjects with clinically significant hematology parameters after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant Clinical Chemistry Laboratory Results
Description: To evaluate the safety by assessing the number of subjects with clinically significant clinical chemistry laboratory results after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Safety of Omega-3-carboxylic Acids by Assessing Number of Subjects With Clinically Significant Urinalysis
Description: To evaluate the safety by assessing the number of subjects with clinically significant urinalysis results after administration of single doses of the omega-3-carboxylic acids test formulations and Epanova in healthy subjects
Time Frame: From screening (within 28 days of first dosing) up to 14 days after last dosing
Population: as for outcome 25
Measure: Number; unit: Participants
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Number analyzed (Participants) | 38 | 39 | 37 | 37 | 39 | 41 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: approximately 12 weeks and Part 2: approximately 10 weeks (i.e. from screening ≤28days until 10-14 days after last dosing).
Description: The safety of subjects were ensured from the pre-defined time points for screening until follow-up (10 to 14 days after last dosing).
Arm/Group | Treatment A_Part 1 | Treatment B_Part 1 | Treatment C_Part 1 | Treatment D_Part 1 | Treatment A_Part 2 | Treatment B_Part 2 | Treatment C_Part 2
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/37 | 0/37 | 0/39 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 8/38 | 7/39 | 4/37 | 5/37 | 3/39 | 3/41 | 3/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A_Part 1 (N=38) | Treatment B_Part 1 (N=39) | Treatment C_Part 1 (N=37) | Treatment D_Part 1 (N=37) | Treatment A_Part 2 (N=39) | Treatment B_Part 2 (N=41) | Treatment C_Part 2 (N=41)
Eyelid Edema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Hyperemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter Site Bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter Site Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel Puncture Site Hematoma (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Catheter Site Phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.